CLINICAL TRIAL: NCT05102097
Title: Effectiveness of Treadmill Walk on Clinical and Functional Variables of Chronic Low Back Pain Patients
Brief Title: Effectiveness of Treadmill Walk on Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayero University Kano, Nigeria (Other)
Responsible Party: Principal Investigator, Rahanatu Abubakar Abba, Principal Investigator, Bayero University Kano, Nigeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPS/18/MPT/00018
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-10

CONDITIONS: Chronic Low Back Pain
Keywords: Treadmill walk
MeSH Terms: interventions — Warm-Up Exercise; Cool-Down Exercise; Standard of Care

STUDY DESIGN:
Intervention Model Description: Group A (experimental group) participants in this group will walk on treadmill and perform standard of care in form of exercises. Group B (Control Group) participants in this group will receive standard of care alone
Who Masked: Outcomes Assessor
Masking Description: Upon completion of baseline assessments, participants will be randomly assigned into two groups A and B in 1:1 ( i.e 20 participants per group) ratio using table of random digit generated from excel.
  The study will be single-blind whereby only the outcome assessors will be blinded to participant's group allocation but the type of intervention will not be specified. Because of the nature of the intervention it will be difficult to blind the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Treadmill walk: i- warm up ( 5 minutes ) II- Main exercise (30 minutes) III- cool down (5 minutes) IV- Standard of care (10minutes)
  Interventions: Behavioral: Warm-up; Behavioral: Main exercise; Behavioral: Cool down; Behavioral: Standard of care
- Control group (Active Comparator): Standard of care (10 minutes)
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Warm-up — Participants will walk on treadmill at a speed of 1.7 mile per hour (MPH) and 0 inclination each session for 6weeks 3 times in a week
  Arms: Experimental Group
Behavioral: Main exercise — Participants will walk on a treadmill with a starting speed of 1.7 mile per hour with inclination of 1 to 4% starting with 1% and increased by 1% each week until 4 weeks and at week 5 and 6 speed will be increased to 5mile per hour starting from 1.7mile per hour and increased by 0.5 mile per hour each 1minute while inclination will be increased to 5% in week 5 and 6% in week 6. Main exercise will be perform 3 times in a week for 6 weeks
  Arms: Experimental Group
Behavioral: Cool down — Participants will walk on treadmill at the speed of 1.7 mile per hour 0 inclination each session for 6 weeks 3 times in a week
  Arms: Experimental Group
Behavioral: Standard of care — Participants will perform Abdominal hollowing, isometric back extension exercise, bridging exercise, graded active flexion, graded active extension by holding for 5seconds and repeated 10times

SUMMARY:
Chronic low back pain is a common health problem with a multifactorial impact on core muscle function as well as causing pain, functional disability and decrease in quality of life, this occur due to the reduction in the physical activity level of the individual causing atrophy and inhibition of the core muscle affecting the stability of the spine

DETAILED DESCRIPTION:
There are several approaches and methods of treating chronic low back pain (CLBP) ranging from education, exercise, electrotherapy and Manual therapy; to alternative treatment such as acupuncture, yoga and Chiropractic. Among the above mention treatment exercise, manual therapy and education are the most frequently utilize for the management of CLBP. The general recommendation for individual with CLBP is to remain active as possible and this can be achieve through exercise.

Evidence shows that active treatment in form of strengthening exercise of the abdominal and back muscles, core stabilization exercise, coordination exercise and aerobic exercise leads to significant reduction in pain and functional disability in patients with CLBP. A number of researches have been focusing on core stability exercise, which is an effective way of recruiting the core muscle (including the abdominal, back, pelvic and hip muscles) that leads to the optimal force production, control of lumbopelvic-hip movement and load transfer from the spine to the pelvis and the lower extremities. The core stabilization exercise has been establish to activate and strength the deep core muscles, but researches are now focusing on the exercise that can be able to activate the core muscles as well as increase the overall health status of the individual

ELIGIBILITY:
Inclusion Criteria:

* male and females between the age of 18 to 65years
* participants attending Usmanu Danfodiyo University teaching Hospital, Sokoto State Specialist Hospital and Orthopedic Hospital
* participants with chronic non-specific low back pain

Exclusion Criteria:

* participants with current low back pain for less than 12 weeks
* participants with cognitive and visual impairment
* participants with other co-morbidities ( systemic disease, carcinomas, organ disease)
* Participants with other neurological findings such as loss of sensation, radiculopathy, parenthesis
* Body mass index of more than 30 Kilogram per meter square
* participants who are pregnant
* participants who had spinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-10-07 (Estimated); Study Completion 2023-01-05 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 5minutes
  A scale of 0 to 10 with 0 indicating no pain and 10 worst pain will be administered to the participants to choose a number indicating their level of pain this will be recorded at base line and 6 weeks after intervention
Electromyograph | 10minutes
  Muscle activity of both lumbar multifidus muscle and rectus abdominous muscle will be assess using neurotrac myoplus pro machine and surface electrode. The assessment will be done both at baseline and at 6weeks after intervention
Biering-sorensen test | 3 minutes
  Participant in prone position stabilize at both ankle and hip with the upper trunk out of the plinth will be instructed to extend the trunk and hold position, the more the time the participant is able to hold the position the more the core muscle endurance
Abdominal dynamic test | 3 minutes
  Participants in supine lying position with the knees flexed to 90 degrees and upper limbs across the chest will be instructed to raised the trunk and neck and hold the position this will be timed using stopwatch. The more the time the participant is able to hold the position the more the core muscle endurance
Flexion rotation test | 3 minutes
  Participants in supine position the knees flex the participants will be instructed to touch alternate knees for 90 seconds and number of repetition will be recorded. The higher the number of repetition the more the core muscle endurance
Pressure biofeedback stabilizer | 4 minutes
  Pressure biofeedback stabilizer will be use to assess the strength of rectus abdominous and Lumbar multifidus muscle strength, the pressure biofeedback stabilizer is a simple device that sense changes in pressure with movement, the pressure cell measures from 0-200millimeter of mercury (mmHg), with a precision of 2 millimeter of mercury with 0 being the lowest score and 200 the highest score. To measure any of the core muscle strength the pressure biofeedback stabilizer will be inflated to 70 millimeter of mercury and will be placed underneath the muscle of the participant and instruction will be giving to the participant to contract the muscle by pressing the inflator down, the reading on the sphygmomanometer will then be recorded.

SECONDARY OUTCOMES:
Oswestry disability index | 10 minutes
  This questionnaire will be administered to the participant both English and hausa version will be use pending on the preference of the participant will be ask to fill so as to know their level of functional disability at baseline and 6 weeks after administration. The questionnaire is scored from 0 indicating no disability and 100 maximum disability
Short form health survey questionnaire | 10 minutes
  Short form health survey questionnaire will be administered to the participants the English or Hausa version pending on the participant preference and their quality of life will be assessed both at baseline and 6weeks intervention. The questionnaire will be scored from 0 to 100, with 0 indicating poor quality of life and 100 highest score in terms of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Rahanatu A Abba, Msc, Principal Investigator — Usmanu Danfodiyo University Teaching Hospital Sokoto, Nigeria
Locations (1):
- Usmanu Danfodiyo University Teaching Hospital Sokoto, Sokoto, Nigeria

IPD SHARING:
Plan to Share IPD: No